CLINICAL TRIAL: NCT01662297
Title: Comparison of Quetiapine and Trazodone Treatment for Insomnia in Dually Diagnosed Veterans: an Open (e.g. Unblinded) Randomized Stay-Switch Pilot Trial
Brief Title: Comparison of Quetiapine and Trazodone Treatment for Insomnia in Dually Diagnosed Veterans
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: it became clear that recruitment was infeasible
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Quetiapine-Trazodone Insomnia; VA MIRB #01579 (Other: VA MIRB #01579)
Record Dates: First submitted 2012-07-16; First posted 2012-08-10 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Insomnia; Mental Health Disorder; Substance Use Disorder
Keywords: Quetiapine; Trazodone; Insomnia; Dual Diagnosis
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mental Disorders; Substance-Related Disorders | interventions — Quetiapine Fumarate; Trazodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine (Active Comparator): Veterans remaining on quetiapine for insomnia.
  Interventions: Drug: Quetiapine
- Trazodone (Active Comparator): Veterans switching from quetiapine to trazodone for the treatment of insomnia.
  Interventions: Drug: Trazodone

INTERVENTIONS:
Drug: Quetiapine — Quetiapine will be administered at a dosage prescribed by veterans' current providers for the treatment of insomnia.
  Other Names: Seroquel; Quetiapine Fumarate
  Arms: Quetiapine
Drug: Trazodone — Veterans willing to switch from quetiapine to trazodone for the treatment of insomnia will receive up to 400mg of trazodone daily.
  Other Names: Desyrel; Oleptro
  Arms: Trazodone

SUMMARY:
This is a pilot comparative effectiveness study designed to determine whether trazodone is as effective as quetiapine for treatment of insomnia in veterans with a history of addiction and mental health issues. The study will have two concurrent phases (parts); first an acceptability determination phase, to determine whether and why (or why not) veterans already taking quetiapine are willing to try an alternative to quetiapine for sleep; and second, a randomized trial phase which will test whether staying on quetiapine has any advantage over switching to trazodone. The purpose of the first phase will be a) to document the proportions of patients and physicians who are willing to agree to such a switch, b) to characterize sociodemographic and clinical characteristics of potentially eligible subjects associated with a willingness to switch from quetiapine to trazodone and c) to record the reasons given why patients and their prescribers are (or are not) willing to accept a switch from quetiapine to trazodone. It will also function to provide some educational background to patients and a reminder to providers about the potential severe side-effects of quetiapine, and will thus facilitate clinical informed consent for the clinical trial phase of the study. Completion of the first part of the study will also serve as the screening component for part II. Part II includes, first, obtaining written informed consent from eligible subjects, and then randomly assigning them to continue quetiapine or to be switched to trazodone in open-label "real world" fashion for the duration of 4 weeks, followed by another four weeks of open, non-randomized follow- up. The purpose of the second part of the study is to determine if trazodone is an adequate substitute for quetiapine, primarily in terms of treating insomnia. The investigators hypothesize that trazodone will not be inferior to quetiapine in maintaining good quality of sleep measured by sleep scales (i.e., scores will not significantly worsen once switched). This study is open to Veterans in the VA system only. Eligible subjects must have a history of "dual diagnosis" (i.e., a history of addiction and mental illness).

DETAILED DESCRIPTION:
Part I of the study involves identification through VA records of subjects eligible for the study based on their prescription of quetiapine. Potentially eligible subjects will be contacted by the research team. Subjects will answer a brief questionnaire about their experience with the medication quetiapine as used for insomnia. If subjects are interested in participated in part II, the clinical trial portion of the study, they will be further screened for eligibility.

Part II consists of a 4 week clinical trial in which subjects are randomized to stay on quetiapine or switch to trazodone, all of which will be open-label. Subjects will be evaluated for symptoms of sleep quality and excessive daytime sleepiness. subjects will also be assessed for changes in mood, and alcohol/drug use. After the initial 4 week treatment period, subjects on trazodone can choose to switch back to quetiapine or continue on trazodone. Subjects will also be evaluated after an additional 4 weeks (8weeks from start of the study) on outcome measures.

ELIGIBILITY:
Inclusion/Exclusion Criteria (PHASE 1):

* Identified by their VA prescribing provider as taking quetiapine primarily as a sedative/hypnotic agent for some form of insomnia for at least 1 month
* Identified by their VA prescribing provider as having dual diagnosis; a lifetime history of substance use disorder and a mental disorder
* Willing to meet with a research assistant to answer several questions regarding their use of and experience with quetiapine.
* Appear not to be regularly on any medication which would be an exclusion for Part II (see Part II exclusion criteria).

Inclusion Criteria (PHASE 2):

* Willing to provide written informed consent.
* Provider reports that primary use of quetiapine is for insomnia for at least one month and not primary or augmentation treatment of mood, anxiety disorder, psychosis, or mood stabilization.
* Have a self-identified and provider confirmed lifetime history of mental health and substance use disorder (dual diagnosis).
* Currently taking Quetiapine up to 300mg daily for the primary purpose of treating insomnia, and have been taking it for at least 1 month (30 days).
* Use of an acceptable method of birth control by female patients who have a possibility of becoming pregnant.
* The provider should review the patients from the identified charts, and fill out information about the patient and why they are on the drug, and provider should consent to us approaching the client and potentially switching them; the investigators will not approach and begin enrollment for part II on subjects if their provider feels it is not appropriate for them for any reason.

Exclusion Criteria (PHASE 2):

* Physiologic substance dependence requiring detoxification in the past 30 days (substance abuse is not an exclusion).
* Concomitant administration of: other sedative hypnotics, benzodiazepines, prazosin, other atypical antipsychotics, stimulants, ketoconazole and other inhibitors of cytochrome P450 3A (e.g., itraconazole, fluconazole, erythromycin, and protease inhibitors), phenytoin or other strong inducers of cytochrome P450 enzymes.
* Intolerance or hypersensitivity to trazodone.
* Pregnant or lactating women or women planning to become pregnant.
* Hepatic or renal problems AST or ALT (>3 times upper limit of normal);
* Elevated bilirubin (>1.2), BUN (>24), creatinine (>1.7).
* Unstable, serious medical condition or one requiring acute medical treatment, or anticipation of hospitalization for extended care.
* Dementia, epilepsy, insulin-dependent diabetes, anticoagulation with coumadin.
* Legal entanglements or pending legal charges with potential of incarceration.
* Recent (i.e., past 3 months) assault or suicide gesture currently needing acute intervention.
* Concurrent participation in another clinical trial with an investigational drug during the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert J Arias, MD, MS, Principal Investigator — Yale University/Veterans Affairs CT; Elizabeth Ralevski, Ph.D., Study Director — Yale University/Veterans Affairs CT
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quetiapine | Trazodone
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine | Trazodone | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] |  | 60 [60 to 60] | 60 [60 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Pittsburgh Sleep Quality Inventory (PSQI)Score
Description: Data analyzed for change from score at baseline, to week 4, to week 8. The range of scores is 0-21 on this scale, with higher scores indicating worse sleep quality. Data will be presented and analyzed for those time points with the main outcome measured as the change from baseline to week 4. This is a comparison between groups (trazodone versus quetiapine)of the change on TOTAL PSQI scores over time using repeated measures analysis. This is a non-superiority analysis, so the hypothesis is that there is no significant difference between treatments. The first four weeks of treatment is the active acute experiment phase, and this will be the main comparison time period for the endpoint, but the investigators will also analyze change in PSQI until the follow-up point at the end of week 8.
Time Frame: From baseline (week 0) to end of 4 week and end of week 8
Population: We had difficulty recruiting and retaining subjects for this study. 3 subjects were randomized and only 1 provided data beyond baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Trazodone
Number analyzed (Participants) | 0 | 1
units on a scale
  change at week 4 |  | -11 (0)
  change at week 8 |  | -11 (0)

2. Secondary Outcome: Change in Insomnia Severity Index (ISI) Scores
Description: THE RANGE OF SCORES IS FROM 0-28, WITH 28 REPRESENTING SEVERE INSOMNIA SYMPTOMS. Measurements made and reported at baseline, week 2, week 4. Data will be presented and analyzed for those time points with the main outcome measured as the change from baseline to week 4. . This is a comparison between groups (trazodone versus quetiapine)of the change on TOTAL ISI scores over time using repeated measures analysis. This is a non-superiority analysis, so the hypothesis is that there is no significant difference between treatments. The investigators will first report the comparison during the active treatment phase (baseline to end of week 4) as the main comparison, but will also examine and report changes on the outcome at the follow up point (end of week 8).
Time Frame: from baseline (week 0) to the end of week 4 and at week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Trazodone
Number analyzed (Participants) | 0 | 1
units on a scale
  change at week 4 |  | -14 (0)
  change at week 8 |  | -16 (0)

3. Secondary Outcome: Change in Epworth Sleepiness Scale (ESS) Over Time
Description: Measurements made at baseline, week 2, week 4, week 8. Data will be presented and analyzed for those time points with the main outcome measured as the change from baseline to week 4. The change from week 4 to week 8 (post-intervention) will also be measured and analyzed, reported. This is a comparison between groups (trazodone versus quetiapine)of the change on ESS scores over time using repeated measures analysis. This is a non-superiority analysis, so the hypothesis is that there is no significant difference between treatments. The investigators will first report the comparison during the active treatment phase (baseline to end of week 4) as the main comparison, but will also examine and report changes on the outcome at the follow up point (end of week 8).The minimum score on ESS is 0-24 units, with higher score representing greater sleepiness.
Time Frame: From baseline (week 0) to end of week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Trazodone
Number analyzed (Participants) | 0 | 1
units on a scale
  change at week 4 |  | -3 (0)
  change at week 8 |  | -4 (0)

4. Secondary Outcome: Change in RAND Short Form 36 Item Health Survey (RAND-SF36) General Health Subscale Over Time
Description: Scores range from 0-100 representing percentage, with a higher score representing better functioning. Measurements made at baseline, week 2, week 4, week 8. Data will be presented and analyzed for those time points with the main outcome measured as the change from baseline to week 4. The change from week 4 to week 8 (post-intervention) will also be measured and analyzed, reported. This is a comparison between groups (trazodone versus quetiapine)of the change on RAND-SF36 scores over time. This is a non-superiority analysis, so the hypothesis is that there is no significant difference between treatments. The investigators will first report the comparison during the active treatment phase (baseline to end of week 4) as the main comparison, but will also examine and report changes on the outcome at the follow up point (end of week 8).
Time Frame: from week 0 (baseline) to end of week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total points possible
Arm/Group | Quetiapine | Trazodone
Number analyzed (Participants) | 0 | 1
percentage of total points possible
  change at week 4 |  | 15 (0)
  change at week 8 |  | 0 (0)

5. Secondary Outcome: Change in Brief Symptom Inventory (BSI) Over Time
Description: The Brief Symptom Inventory scale measures a broad range of psychiatric symptoms (psychological distress) and is meant to provide an overall measure of mental health symptomatology. The BSI has 53 items that use a 5-item Likert scale response. In general, higher scores correspond to greater symptomatology and distress. Usually, the range of scores goes from 0 - 4, since it is averaged over the number of responses, however, we report the raw total score which is the sum of all responses, thus the range is 0-212. Measurements made at baseline, week 2, week 4, week 8. Data will be presented and analyzed for those time points with the main outcome measured as the change from baseline to week 4. This is a comparison between groups of the change on BSI scores over time using repeated measures analysis. This is a non-superiority analysis, so the hypothesis is that there is no significant difference between treatments.
Time Frame: from week 0 (baseline) to end of week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Trazodone
Number analyzed (Participants) | 0 | 1
units on a scale
  change at week 4 |  | -48
  change at week 8 |  | -48

6. Secondary Outcome: Change in Alcohol Urge Questionnaire (AUQ)Scores Over Time
Description: The lowest possible score for the AUQ is 8 (representing less urge to drink) and the highest score would be a 56 (more urge to drink). Measurements made at baseline, week 2, week 4, week 8. Data will be presented and analyzed for those time points with the main outcome measured as the change from baseline to week 4. This is a comparison between groups (trazodone versus quetiapine)of the change on AUQ scores over time. This is a non-superiority analysis, so the hypothesis is that there is no significant difference between treatments. The investigators will first report the comparison during the active treatment phase (baseline to end of week 4) as the main comparison, but will also examine and report changes on the outcome at the follow up point (end of week 8).
Time Frame: from week 0 (baseline) to end of week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Trazodone
Number analyzed (Participants) | 0 | 1
units on a scale
  change after week 4 |  | -1 (0)
  change after week 8 |  | -12 (0)

7. Secondary Outcome: Percentage of Heavy Drinking Days
Description: This is a comparison between groups of the mean percent heavy drinking days during the first 4 weeks, and then through to the follow up point (end of week 8). The investigators will first report the comparison during the active treatment phase (baseline to end of week 4) as the main comparison, but will also examine and report changes on the outcome at the follow up point (end of week 8).
Time Frame: from week 0 (baseline) to end of week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Quetiapine | Trazodone
Number analyzed (Participants) | 0 | 1
percentage of heavy drinking days
  percentage at week 4 |  | 0 (0)
  percentage at week 8 |  | 0 (0)

8. Secondary Outcome: Percentage of Negative Urine Drug Screens
Description: This is a comparison between groups of the mean percent of negative urine drug screens. The investigators will first report the comparison during the active treatment phase (baseline to end of week 4) as the main comparison, but will also examine and report changes on the outcome at the follow up point (end of week 8). THIS IS A CUMULATIVE PERCENTAGE. MAXIMUM SCORE IS 100%, MINIMUM 0%.
Time Frame: from week 0 (baseline) to end of week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of tests
Arm/Group | Quetiapine | Trazodone
Number analyzed (Participants) | 0 | 1
percentage of tests
  cumulative percentage at week 4 |  | 0 (0)
  cumulative percentage at week 8 |  | 0 (0)

9. Secondary Outcome: Medical Outcomes Study Sleep Scale- Sleep Index (Short)
Description: THE RANGE OF SCORES IS FROM 0-100, WITH 100 REPRESENTING SEVERE INSOMNIA SYMPTOMS. Measurements made and reported at baseline, week 2, week 4. Data will be presented and analyzed for those time points with the main outcome measured as the change from baseline to week 4. . This is a comparison between groups (trazodone versus quetiapine)of the change on TOTAL MOS-SS scores over time using repeated measures analysis. This is a non-superiority analysis, so the hypothesis is that there is no significant difference between treatments. The investigators will first report the comparison during the active treatment phase (baseline to end of week 4) as the main comparison, but will also examine and report changes on the outcome at the follow up point (end of week 8).
Time Frame: from baseline (week 0) to the end of week 8 sample
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Trazodone
Number analyzed (Participants) | 0 | 1
units on a scale
  change at 4 weeks |  | -13.33 (0)
  change at 8 weeks |  | -26.66 (0)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Quetiapine | Trazodone
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine (N=0) | Trazodone (N=1)
Death (Cardiac disorders) | 0 (0) | 1 (1) — This patient died after completing the study and the 8 week follow up session. Subject died on 4/30/2013, several weeks after completing the follow up period for the study (4/8/13). The death was clearly unrelated to study participation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine (N=0) | Trazodone (N=1)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No